CLINICAL TRIAL: NCT05333523
Title: Personalized Elective Neck Irradiation Guided by Sentinel Lymph Node Biopsy in Patients With Squamous Cell Carcinoma of the Oropharynx, Larynx or Hypopharynx With a Clinically Negative Neck: (Chemo)Radiotherapy to the PRIMary Tumor Only. The PRIMO Study.
Brief Title: Personalized Elective Neck Irradiation Guided by Sentinel Lymph Node Biopsy in Larynx and Pharynx Cancer. The PRIMO Study.
Acronym: PRIMO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: UMC Utrecht (Other); The Netherlands Cancer Institute (Other); Erasmus Medical Center (Other); Leiden University Medical Center (Other); Maastro Clinic, The Netherlands (Other); Maastricht University Medical Center (Other); University Medical Center Groningen (Other); Radiotherapiegroep (Other); Rijnstate Hospital (Other); Medisch Spectrum Twente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRIMO v2.0 dd20250401
Record Dates: First submitted 2022-03-31; First posted 2022-04-19 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Laryngeal Squamous Cell Carcinoma; Hypopharynx Squamous Cell Carcinoma; Oropharyngeal Squamous Cell Carcinoma
Keywords: Head and neck cancer; Squamous cell carcinoma; Sentinel lymph node biopsy; Elective neck irradiation; FDG-PET
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sentinel lymph node biopsy guided selective elective neck irradiation (Experimental): * Sentinel lymph node biopsy
  * Radiotherapy (IMRT/VMAT with SIB) to the primary tumor with selective elective neck irradiation guided by histopathologic status of the sentinel lymph node(s)
  Interventions: Radiation: Sentinel lymph node biopsy guided selective elective neck irradiation
- Standard elective neck irradiation (Active Comparator): - Radiotherapy (IMRT/VMAT with SIB) to the primary tumor with standard bilateral elective neck irradiation
  Interventions: Radiation: Standard elective neck irradiation

INTERVENTIONS:
Radiation: Sentinel lymph node biopsy guided selective elective neck irradiation — Patients will undergo sentinel lymph node biopsy. Based on the histopathologic status of the sentinel lymph node(s), selective elective neck irradiation is performed with standard radiation treatment of the primary tumor.
  There are 3 possible treatment scenarios.
  1. Bilateral elective neck irradiation is indicated when lymph nodes at both sides of the neck contain metastases or when sentinel lymph node detection fails.
  2. Unilateral elective neck irradiation is indicated when lymph nodes at one side of the neck only contain metastases.
  3. Full omission of elective neck irradiation is indicated when lymph nodes at both sides of the neck are free of metastases.
  Arms: Sentinel lymph node biopsy guided selective elective neck irradiation
Radiation: Standard elective neck irradiation — Patients randomized to the control arm will receive the standard of care, according to (inter)national clinical practice guidelines. This will consist of (chemo)radiotherapy to the primary tumor with standard elective neck irradiation in all patients. No sentinel lymph node biopsy will be performed.
  Arms: Standard elective neck irradiation

SUMMARY:
Rationale | Elective neck irradiation is performed in head and neck cancer patients treated with definitive (chemo)radiotherapy. The aim is to eradicate nodal metastases that are not detectable by pretreatment imaging techniques. It is conceivable that personalized neck irradiation can be performed guided by the results of sentinel lymph node biopsy. It is expected that elective neck irradiation can be omitted to one or both sides of the neck in 9 out of 10 patients with a clinically negative neck (cN0). For patients with clinically positive ipsilateral nodes (cN1-2b), it is expected that elective irradiation of the contralateral neck can be omitted in 7 out of 10 patients. This will enable better sparing of normal tissues from radiation and result in less permanent long-term radiation side effects with better quality of life.

Methods/design | This is a multicenter randomized controlled trial aiming to compare safety and efficacy of treatment with sentinel lymph node biopsy guided neck irradiation versus standard bilateral elective neck irradiation in 242 patients with cN0-N2b squamous cell carcinoma of the oropharynx, larynx or hypopharynx for whom bilateral elective neck irradiation is indicated. Patients randomized to the experimental-arm will undergo sentinel lymph node biopsy. Based on the histopathologic status of the sentinel lymph nodes, patients will receive no elective neck irradiation (if no nodal metastases found at both sides of the neck), unilateral neck irradiation only (if no nodal metastases found at contralateral side of the neck only) or bilateral neck irradiation (if nodal metastases found at both sides of the neck). Patients randomized to the control arm will not undergo sentinel lymph node biopsy but will receive standard bilateral elective neck irradiation. The primary safety endpoint is the number of patients with recurrence in regional lymph nodes within 2 years after treatment. The primary efficacy endpoint is patient reported xerostomia-related quality of life at 6 months after treatment.

Discussion | If this trial demonstrates that the experimental treatment is non-inferior to the standard treatment in terms of regional recurrence and is superior in terms of xerostomia-related quality of life, this will become the new standard of care.

DETAILED DESCRIPTION:
Rationale | Squamous cell carcinoma of the upper aerodigestive tract comes with a substantial risk for cervical lymph node metastases. Elective neck irradiation is performed in patients receiving (chemo)radiotherapy aiming to eradicate eventual nodal metastases that are under the detection level of pretreatment imaging techniques. Most toxicity and permanent long-term radiation side effects are caused by elective neck irradiation. In particular xerostomia and dysphagia are notoriously known to negatively and permanently affect quality of life. Sentinel lymph node biopsy has emerged as a staging procedure that can reliably detect microscopic metastases by histopathological examination of sentinel lymph nodes and the pathologic status of the sentinel lymph node accurately reflects the status of the remaining nodal basin. A recent meta-analysis demonstrated an excellent diagnostic test accuracy of sentinel lymph node biopsy in patients with cancer of the oropharynx, larynx and hypopharynx (sensitivity 0.93 and negative predictive value 0.97). It is conceivable that personalized neck irradiation can be performed guided by the results of sentinel lymph node biopsy. With this approach it is expected that elective neck irradiation can be omitted to one or both sides of the neck in 9 out of 10 patients with a clinically negative neck (cN0). For patients with clinically positive ipsilateral nodes (cN1-2b), it is expected that elective irradiation of the contralateral neck can be omitted in 7 out of 10 patients. This will enable better sparing of normal tissues from radiation and result in less permanent long-term radiation side effects with better quality of life.

Objective | To compare safety and efficacy of treatment with sentinel lymph node biopsy guided neck irradiation versus standard elective neck irradiation in patients receiving definitive (chemo)radiotherapy for squamous cell carcinoma of the oropharynx, larynx or hypopharynx.

Design | This is a multicenter, randomized controlled trial. In total 242 patients will be randomized in ratio 1:1 to the control arm with standard bilateral elective neck irradiation or to the interventional arm with sentinel lymph node biopsy guided neck irradiation. During a 2 year follow-up, data on toxicity, quality of life and oncologic outcomes will be collected. If this trial demonstrates that the interventional treatment is non-inferior to the standard treatment in terms of regional recurrence and is superior in terms of xerostomia-related quality of life, this will become the standard of care.

Population | Patients to be treated with definitive (chemo)radiotherapy for stage cT1-4N0-2bM0 squamous cell carcinoma of the oropharynx, larynx or hypopharynx for whom bilateral elective neck irradiation is indicated. Excluded are patients with recurrent disease or patients who received previous oncologic surgery or radiotherapy to the neck.

Intervention | Patients randomized to the intervention arm will undergo sentinel lymph node biopsy. For patients with a clinically negative neck (cN0), sentinel lymph node biopsy is performed bilaterally. Based on the histopathologic status of the sentinel lymph node(s), patients will receive no elective neck irradiation (if all sentinel lymph nodes are negative), unilateral neck irradiation only (if a sentinel lymph node is positive at one side of the neck) or bilateral neck irradiation (if sentinel lymph nodes are positive at both sides of the neck). For patients with clinically positive ipsilateral nodes (cN1-2b), sentinel lymph node biopsy is performed contralaterally only. Contralateral elective neck irradiation will only be performed when sentinel lymph nodes are positive. For patients randomized to the control arm sentinel lymph node biopsy will not be performed and all will receive standard bilateral elective neck irradiation (with boost to clinically positive ipsilateral nodes (cN1-2b) if present).

Primary endpoints | The primary safety endpoint is the number of patients with recurrence in regional lymph nodes (in the absence of synchronous recurrence of the primary tumor, or initially clinically positive nodes, or second primary tumor) within 2 years after treatment. The primary efficacy endpoint is patient reported xerostomia-related quality of life measured by the xerostomia symptom scale of the EORTC QLQ-H&N35 at 6 months after treatment.

Other endpoints | Acute and late radiation toxicity, quality of life after treatment with focus on xerostomia and dysphagia, local and regional control rates, disease specific and overall survival, and cost-effectiveness.

Burden associated with participation | Patients randomized to the intervention arm will undergo sentinel lymph node biopsy (flexible endoscopic tracer injection under topical anesthesia in the outpatient clinic, SPECT/CT-scan and surgical removal of identified sentinel lymph nodes under general anesthesia). These procedures will not be performed in patients in the control arm. For patients randomized to the intervention arm there is a potential increased risk for regional recurrence because elective neck irradiation is omitted based on the histopathologic status of the sentinel lymph node(s). However this risk is expected to be very small (3.1% versus 2.0% in the control arm). Because regional recurrences can be cured in 70-90% of the patients with salvage neck dissection, the effect on overall survival is expected to be negligible. Independent of randomization, participants will undergo non-invasive procedures to objectify radiation sequelae and will be asked to complete quality of life questionnaires.

Benefit associated with participation | With sentinel lymph node biopsy, it is expected that futile elective neck irradiation can be omitted to one or both sides of the neck in most patients. This will enable better sparing of normal tissues from radiation and it is expected that this will result in a major decrease of permanent long-term radiation side effects (such as xerostomia and dysphagia) with better quality of life after treatment compared to standard elective neck irradiation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) with newly diagnosed cT1-4N0-2bM0 squamous cell carcinoma of the oropharynx (HPV-), larynx or hypopharynx, or cT1-4N0-1M0 oropharynx (HPV+) (AJCC TNM 8)
* Histopathological diagnosis of squamous cell carcinoma.
* Adequate staging of the neck including CT or MRI, and 18F-FDG-PET demonstrating no contralateral lymph node metastases.
* Recommendation for curative intent external beam (chemo)radiotherapy made by a multidisciplinary head and neck oncology team (in case of chemoradiotherapy, only patients receiving concomitant platinum-based regimen are eligible).
* Bilateral ENI is indicated according to Dutch consensus guidelines (LPHHRT) (see Appendix 13.1).
* Procedures for SLNB (i.e. tumor accessible for tracer injection, imaging and surgery under general anesthesia) are deemed feasible by the head and neck surgeon.

Exclusion Criteria:

* Recurrent disease or previous anticancer treatment to the head and neck area (e.g. radical attempt or tumor reductive surgery, neck dissection, neo-adjuvant chemotherapy or radiotherapy) except for endoscopic glottic laser micro surgery.
* Well lateralized oropharyngeal cancers and early stage laryngeal cancers requiring no or unilateral ENI according to Dutch consensus guidelines (LPHHRT)
* Patients receiving concomitant non-platinum-based systemic agents (e.g. cetuximab).
* Patients that qualify for proton therapy and want to be treated accordingly.
* Compromised airway or tracheostomy.
* Any active invasive malignancy within the last 3 years except for early stage basal/squamous cell carcinoma of the skin and incidental finding of stage T1N0M0 prostate cancer.
* Any somatic, psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol or follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2029-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with regional recurrence | 24 months
  Only recurrence in regional lymph nodes in the absence of synchronous recurrence of the primary tumor or initially clinically positive nodes, or second primary head and neck tumors are considered as events
Patiënt reported xerostomia related quality of life as assessed by EORTC Quality of Life Questionnaire Head and Neck Module (QLQ-H&N35) | 6 months

CONTACTS AND LOCATIONS:
Locations (9):
- Netherlands (9):
  - The Netherlands Cancer Institute, Amsterdam
  - Radiotherapiegroep / Rijnstate Ziekenhuis, Arnhem
  - Medisch Spectrum Twente (MST), Enschede
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - MAASTRO Clinic / Maastricht University Medical Center, Maastricht
  - Radboud University Nijmegen Medical Center, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - University Medical Center Utrecht, Utrecht

REFERENCES:
- [Background] van den Bosch S, Takes RP, de Ridder M, de Bree R, Al-Mamgani A, Schreuder WH, Hoebers FJP, van Weert S, Elbers JBW, Hardillo JA, Meijer TWH, Plaat BEC, de Jong MA, Jansen JC, Wellenstein DJ, van den Broek GB, Vogel WV, Arens AIJ, Kaanders JHAM. Personalized neck irradiation guided by sentinel lymph node biopsy in patients with squamous cell carcinoma of the oropharynx, larynx or hypopharynx with a clinically negative neck: (Chemo)radiotherapy to the PRIMary tumor only. Protocol of the PRIMO study. Clin Transl Radiat Oncol. 2023 Oct 26;44:100696. doi: 10.1016/j.ctro.2023.100696. eCollection 2024 Jan. PMID 37965060
- [Background] van den Bosch S, Czerwinski M, Govers T, Takes RP, de Bree R, Al-Mamgani A, Hannink G, Kaanders JHAM. Diagnostic test accuracy of sentinel lymph node biopsy in squamous cell carcinoma of the oropharynx, larynx, and hypopharynx: A systematic review and meta-analysis. Head Neck. 2022 Nov;44(11):2621-2632. doi: 10.1002/hed.27175. Epub 2022 Sep 1. PMID 36047597